CLINICAL TRIAL: NCT06619860
Title: A Phase 2, Randomized, Double-blind, Active-controlled, Dose-ranging, Parallel-design Study of the Efficacy and Safety of Oral VX-993 in Subjects With Pain Associated With Diabetic Peripheral Neuropathy
Brief Title: Evaluation of Efficacy and Safety of VX-993 for Pain Associated With Diabetic Peripheral Neuropathy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX24-993-103; 2024-514689-38-01 (Other: EU Trial (CTIS) Number)
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-04

CONDITIONS: Diabetic Peripheral Neuropathic Pain
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VX-993 (Experimental): Participants will be randomized to receive multiple doses of different dose levels of VX-993.
  Interventions: Drug: VX-993; Drug: Placebo (matched to pregabalin)
- Pregabalin (Active Comparator): Participants will be randomized to receive Pregabalin.
  Interventions: Drug: Pregabalin; Drug: Placebo (matched to VX-993)

INTERVENTIONS:
Drug: VX-993 — Tablets for oral administration.
  Arms: VX-993
Drug: Pregabalin — Capsules for oral administration.
  Arms: Pregabalin
Drug: Placebo (matched to pregabalin) — Placebo matched to pregabalin for oral administration.
  Arms: VX-993
Drug: Placebo (matched to VX-993) — Placebo matched to VX-993 for oral administration.
  Arms: Pregabalin

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of VX-993 in participants with pain associated with Diabetic Peripheral Neuropathy (DPN)

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of diabetes mellitus type 1 or type 2 with

  * Glycosylated hemoglobin A1c (HbA1c) less than or equal to (≤) 9% and
  * Presence of bilateral pain in lower extremities due to DPN (defined as a symmetric, length-dependent sensory or sensorimotor polyneuropathy) for at least 1 year

Key Exclusion Criteria:

* Painful neuropathy other than DPN
* History of cardiac dysrhythmias requiring anti-arrhythmia treatment(s)
* History of a clinical atherosclerotic event, such as myocardial infarction or stroke, within the past 12 months

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in the Weekly Average of Daily Pain Intensity on the Numeric Pain Rating Scale (NPRS) at Week 12 | From Baseline up to Week 12

SECONDARY OUTCOMES:
Proportion of Participants with Greater than or Equal to (≥) 30 Percent (%) Reduction From Baseline in the Weekly Average of Daily Pain Intensity on the NPRS at Week 12 | From Baseline up to Week 12
Proportion of Participants with ≥50% Reduction From Baseline in the Weekly Average of Daily Pain Intensity on the NPRS at Week 12 | From Baseline up to Week 12
Proportion of Participants with ≥70% Reduction From Baseline in the Weekly Average of Daily Pain Intensity on the NPRS at Week 12 | From Baseline up to Week 12
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 up to Week 16

CONTACTS AND LOCATIONS:
Locations (47):
- United States (25):
  - Cullman Clinical Trials, Cullman, Alabama
  - Trovare Clinical Research - Bakersfield CA, Bakersfield, California
  - Eximia Research - San Diego, La Mesa, California
  - Paradigm Clincial Research Centers, LLC., Wheat Ridge, Wheat Ridge, Colorado
  - Accel Research - Deland, DeLand, Florida
  - AMR Fort Myers (The Clinical Study Center), Fort Myers, Florida
  - Velocity Clinical Research - Hallandale Beach, Hallandale, Florida
  - Health Awareness, Inc., Jupiter, Jupiter, Florida
  - Suncoast Research Associates - Miami, Miami, Florida
  - Innovation Medical Research Center - Palmetto, Palmetto Bay, Florida
  - Health Awareness, Inc. - Port St. Lucie, Port Saint Lucie, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Accel Research - Decatur, Decatur, Georgia
  - Velocity Clinical Research - Boise, Meridian, Idaho
  - Healthcare Research Network - Flossmoor IL, Flossmoor, Illinois
  - Quest Research Institute, Farmington Hills, Michigan
  - Healthcare Research Network - Hazelwood MO, Hazelwood, Missouri
  - Eximia Research - Raleigh, Raleigh, North Carolina
  - Velocity Clinical Research - Cleveland, Beachwood, Ohio
  - Velocity Clinical Research - Providence, East Greenwich, Rhode Island
  - Clinical Trials of South Carolina - Berkeley - Moncks Corner, Moncks Corner, South Carolina
  - Gadolin Research, Beaumont, Texas
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - San Antonio Clinical Trials, San Antonio, Texas
  - AMR Norfolk, Norfolk, Virginia
- Canada (4):
  - Centricity Research Brampton, Brampton
  - OCT Research ULC, Kelowna
  - Altasciences - Beaumont Clinic Montreal, Montreal
  - Mount Sinai Hospital - Leadership Sinai Centre for Diabetes (LSCD), Toronto
- France (4):
  - Centre Hospitalier Universitaire de Clermont-Ferrand - Site Gabriel-Montpied, Clermont-Ferrand
  - CHU de Nîmes - Pain Assessment and Treatment Center, Nîmes
  - Hopital Cochin - Rheumatology, Paris
  - North Hospital, Saint-Priest-en-Jarez
- Germany (3):
  - Ruhr-Universitaet Bochum - Heart and Diabetes Center, Bad Oeynhausen
  - FutureMeds GmbH, Berlin
  - FutureMeds Frankfurt, Offenbach/Main
- Italy (2):
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - IRCCS Ospedale San Raffaele - InSpe and Division of Neuroscience, Milan
- United Kingdom (9):
  - Birmingham Heartlands Hospital - Heartlands Hospital Diabetes Centre and MIDRU, Birmingham
  - FutureMeds Birmingham, Birmingham
  - Ninewells Hospital - Endocrinology, Dundee
  - FutureMeds Glasgow, Glasgow
  - University of Liverpool - Aintree University Hospital, Liverpool
  - St Pancras Clinical Research, London
  - Manchester Diabetes Centre (MDC), Manchester
  - George Eliot Hospital NHS Trust, Nuneaton
  - Royal Hallamshire Hospital - Endocrinology, Sheffield

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/